CLINICAL TRIAL: NCT02469506
Title: The Effects of Daily Neuromuscular Electrical Stimulation on Muscle Mass During Long-term Unilateral Ankle Immobilization in Adults With Ankle Fractures
Brief Title: Neuromuscular Electrical Stimulation During Immobilization Due to Ankle Fractures
Acronym: ANKL-ES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Minimal to no inclusion.
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Prof. Dr. Luc. J.C. van Loon, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: METC 14-3-050
Record Dates: First submitted 2015-06-04; First posted 2015-06-11 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Immobilization; Muscle Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NMES group (Experimental): Patients will receive twice daily sessions of neuromuscular electrical stimulation (NMES).
  Interventions: Device: Neuromuscular Electrical Stimulation (NMES)
- Control group (No Intervention): Patients will receive daily visits by the investigator to check progress.

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation (NMES) — The protocol will consist of a warm-up period (5 min), a stimulation period (30min), and a cooling-down period (5min). Stimulation will be provided by an Enraf Nonius TensMed S84 stimulation device.
  Arms: NMES group

SUMMARY:
Rationale: Situations such as fractures of the lower extremity can necessitate a prolonged period of immobilization in otherwise healthy individuals. Long-term immobilization of the lower extremity has shown to cause significant reductions in skeletal muscle mass, already occurring during the early stages of disuse. Accordingly, feasible strategies for attenuating this loss of muscle during disuse need to be pursued. Local neuromuscular electrical stimulation (NMES) offers such a potential strategy but, as yet, remains untested during prolonged muscle disuse in a clinical setting.

Objective: To investigate whether twice daily local (gastrocnemius/soleus) NMES attenuates muscle loss during 2 weeks of unilateral ankle immobilization.

Study design: Randomized, parallel (two groups) study design.

Study population: 30 adults (18-65 y) with any form of closed ankle fractures needing surgical treatment.

Intervention: Twice daily neuromuscular electrical stimulation (NMES) or no intervention.

Main study parameters/endpoints: Primary: Calf muscle (gastrocnemius) cross sectional area (CSA) as determined by CT scan. Secondary: type I and II muscle fiber CSA and SC content, intramuscular triglyceride content and mRNA and protein expression of anabolic signaling proteins.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral closed ankle fracture (Weber type A, B or C)
* Aged from 18-65 years
* 18.5 < BMI < 30 kg/m2
* Undergoing surgical treatment

Exclusion Criteria:

* Additional fractures beside ankle fracture (e.g. multi-trauma following a car accident)
* Use of oral anticoagulants such as vitamin K-antagonists (e.g. acenocoumarol and fenprocoumon) and direct-acting or new oral anticoagulants (e.g. apixaban, dabigatran and rivaroxaban).
* Any family history of thrombosis
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Myocardial infarction within the last 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage change in calf muscle cross sectional area | Baseline measurements will be performed at the day of the surgical intervention for the ankle fracture. Post measurements will be performed at the last day of the subsequent 2-week period of immobilization with a lower leg cast.
  Measured by a single slice CT-scan of the calf muscle.

SECONDARY OUTCOMES:
Percentage change in type I and II muscle fiber cross sectional area | Baseline measurements will be performed at the day of the surgical intervention for the ankle fracture. Post measurements will be performed at the last day of the subsequent 2-week period of immobilization with a lower leg cast.
  Measured by immunohistochemical analyses of the muscle biopsies.
Percentage change in type I and II muscle fiber satellite cell content | Baseline measurements will be performed at the day of the surgical intervention for the ankle fracture. Post measurements will be performed at the last day of the subsequent 2-week period of immobilization with a lower leg cast.
  Measured by immunohistochemical analyses of the muscle biopsies.
Percentage change in type I and II muscle fiber intramuscular triglyceride content | Baseline measurements will be performed at the day of the surgical intervention for the ankle fracture. Post measurements will be performed at the last day of the subsequent 2-week period of immobilization with a lower leg cast.
  Measured by immunohistochemical analyses of the muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Prof, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands